CLINICAL TRIAL: NCT05567770
Title: ACTInium-J591 Radionuclide Therapy in PSMA-Detected Metastatic HOrmone-Sensitive Recurrent Prostate CaNcer
Acronym: ACTION
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Stakeholder elected not to proceed with the study
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Convergent Therapeutics, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-08025155
Record Dates: First submitted 2022-10-03; First posted 2022-10-05 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Prostate Cancer Metastatic
MeSH Terms: interventions — Radiosurgery; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Active Comparator)
  Interventions: Drug: Actinium-J591; Radiation: Stereotactic Body Radiation Therapy
- Cohort 2 (Active Comparator)
  Interventions: Drug: Actinium-J591; Drug: Androgen Deprivation Therapy

INTERVENTIONS:
Drug: Actinium-J591 — Cohort 1 with oligometastatic disease will receive Actinium-J591 and Stereotactic Body Radiation Therapy
Radiation: Stereotactic Body Radiation Therapy — Cohort 1 patients with oligometastatic disease will receive Actinium-J591 and Stereotactic Body Radiation Therapy
  Other Names: SBRT
  Arms: Cohort 1
Drug: Androgen Deprivation Therapy — Cohort 2 patient with Polymetastatic disease will receive Actinium-J591 and Androgen Deprivation therapy (ADT)
  Other Names: ADT
  Arms: Cohort 2

SUMMARY:
The purpose of this study is to evaluate the safety of combining Actinium- J591 with radiation therapy or with androgen deprivation therapy.

DETAILED DESCRIPTION:
This is a two cohort pilot study for patients with hormone-sensitive prostate cancer after primary treatment +/- salvage treatment with metastases detected on PSMA-PET scan but equivocal, indeterminate or absent on conventional imaging.

Cohort 1 will have patients with Oligometastatic (low volume, between 1 and 5 metastases) disease and Cohort 2 will have patients with polymetastatic (high volume, ≥5 metastases) disease detected via PSMA PET.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of prostate adenocarcinoma at any anatomical location (for example, prostate, metastatic site), including intraductal or ductal carcinoma, at any time before registration.
* Age ≥ 18 years
* ECOG Performance Status 0-2.
* Prior curative-intent treatment to the prostate, by either:
* External beam and/or brachytherapy to: Prostate alone, prostate and seminal vesicles, prostate and pelvic nodes, or radiation to all three sites.
* Radical prostatectomy alone, radical prostatectomy plus postoperative radiotherapy to the prostate bed, or radical prostatectomy plus postoperative radiotherapy to the pelvic nodes.
* Must meet study entry criteria based on the following diagnostic workup within 120 days prior to enrollment: • History and physical examination
* 99mTc bone scan (Must be negative or equivocal);
* Either CT or MRI of pelvis +/- abdomen (Must be negative or equivocal);
* PSMA PET scan (Must be positive with exception of local disease); Note: All 3 scans are mandatory (bone scan; CT/MR; PET)
* Serum total testosterone >100 ng/dL within 120 days prior to enrollment.
* Be willing to use effective contraception during the entire study period.
* To have adequate organ and marrow function, as defined below:
* a. Absolute neutrophil count (ANC) of ≥2,000/mm3
* b. Hemoglobin ≥9 g/dL without need for transfusion
* c. Platelet count ≥150,000/mm3 and absent history or primary quantitative or qualitative platelet defect
* d. Serum creatinine of ≤1.5 x ULN or calculated creatinine clearance of ≥60 mL/min/1.73 m2 by Cockcroft-Gault (or determined by 24 hour urine collection)
* e. Serum total bilirubin ≤1.5 x ULN (unless due to Gilbert's syndrome, in which case direct bilirubin must be normal)
* f. Serum AST and ALT ≤1.5 x ULN.

Exclusion Criteria:

* 1. Currently on androgen deprivation or anti-androgen therapy.
* Definitive radiologic evidence of metastatic disease on conventional imaging, defined by one of the following:
* a. osseous metastasis on 99mTc radionuclide bone scan, or
* b. extra pelvic nodal/soft tissue disease (> 1.5cm in short axis) on CT or MRI pelvis +/- abdomen
* Spinal cord compression, or spinal intramedullary, brain, and/or visceral (for example liver, lung, etc.) metastasis. Note: Spinal metastases (PSMA PET- detected) with epidural extension are eligible if there is >0.3cm spatial separation between the gross tumor volume and spinal cord.
* Biopsy-proven prostatic carcinoma with signet-ring, sarcomatoid, or neuroendocrine features (for example, small cell).
* Prior metastatic or non-metastatic, invasive malignancy (except non metastatic, non-melanomatous skin cancer) unless continuously disease free for > 3 years.
* Prior chemotherapy for prostate cancer or bilateral orchiectomy. Note: Prior chemotherapy for a different cancer is allowed if continuously disease-free for > 3 years.
* Intrapelvic lymph nodes as only site of prostate cancer recurrence.
* Received a platelet transfusion within 4 weeks of treatment
* Received growth factors for white blood cells or platelets within 4 weeks of treatment
* Prior treatment with unsealed radiation sources such as 89Strontium or 153Samarium-containing compounds (e.g. Metastron, Quadramet)
* History of prior PSMA-TRT
* Known history of myelodysplastic syndrome
* Other serious illness(es) involving the cardiac, respiratory, central nervous, renal, hepatic, or hematological systems which might preclude completion of this study or interfere with determination of causality of any adverse effects experienced in this study.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) Rate | 24 months
  A DLT will is defined as a grade 3 or higher hematologic adverse event or a grade 2 or higher non-hematologic adverse event deemed to be at least possibly related to study treatment. Adverse events will be assessed using CTCAE version 5. Patients will be observed for a DLT for 3 months from the second dose of actinium-J591.
Change in Maximum Tolerated Dose (MTD) | 3,6,12,18 and 24 months.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) on conventional Imaging | 3 months
Progression Free Survival (PFS) on conventional Imaging | 6 months
Progression Free Survival (PFS) on conventional Imaging | 12 months
Progression Free Survival (PFS) on conventional Imaging | 24 months
Progression Free Survival (PFS) on prostate-specific membrane antigen (PSMA) positron emission tomography (PET) imaging. | 3 months
Progression Free Survival (PFS) on prostate-specific membrane antigen (PSMA) positron emission tomography (PET) imaging. | 6 months
Progression Free Survival (PFS) on prostate-specific membrane antigen (PSMA) positron emission tomography (PET) imaging. | 12 months
Progression Free Survival (PFS) on prostate-specific membrane antigen (PSMA) positron emission tomography (PET) imaging. | 24 months
Changes in PSMA expression measured by comparison of SUV on PSMA PET scans before and after treatment | 3, 6, 12, and 24 months
Change in Percentage of PSA decline | 3, 6, 12, 15, 18, 21, and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Himanshu Nagar, M.D., Principal Investigator — Weill Medical College of Cornell University

IPD SHARING:
Plan to Share IPD: No